CLINICAL TRIAL: NCT06436664
Title: Evaluation of the Effects of Different Tooth Brushing Explanations on Oral Hygiene in Patients With Fixed Orthodontic Treatment
Brief Title: The Effects of Different Tooth Brushing Explanations in Fixed Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Yasemin Tunca, PhD, DDS, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024/01-04
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Orthodontic Treatment; Dental Plaque Induced Gingival Disease
Keywords: tooth brushing; fixed orthodontic treatment; microbial dental plaque
MeSH Terms: interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Other): In patients receiving fixed orthodontic treatment, the orthodontic plaque index, Turesky modified index and gingival index will be recorded at the beginning, 1st and 3rd months. No special instructions will be given to these patients regarding the tooth brushing process.
  Interventions: Other: Tooth brushing
- Group 1 (Experimental): Patients will receive a standard brochure and oral presentation on tooth brushing in the Group 1. The orthodontic plaque index, Turesky modified index and gingival index will be recorded at the beginning, 1st and 3rd months. These patients will receive a standardized brochure for tooth brushing.
  Interventions: Other: Tooth brushing
- Group 2 (Experimental): Patients will receive a standard tooth brushing on a dental model in the Group 2. The orthodontic plaque index, Turesky modified index and gingival index will be recorded at the beginning, 1st and 3rd months.
  Interventions: Other: Tooth brushing
- Group 3 (Experimental): In patients undergoing fixed orthodontic treatment, the orthodontic plaque index, Turesky modified index and gingival index will be recorded at the beginning, 1st and 3rd months. Patients will be taught standard tooth brushing with a video in Group 3.
  Interventions: Other: Tooth brushing

INTERVENTIONS:
Other: Tooth brushing — Firstly, the toothbrush must be positioned at a 45° angle to the gingival margin. Secondly, the brush should be moved back and forth in small horizontal jerks. Thirdly, with a vertical movement, the brush should be moved in the occlusal direction, i.e. upwards in the lower jaw and downwards in the upper jaw to remove debris.

SUMMARY:
The aim of this study is to investigate the effects of tooth brushing training methods on orthodontic patients and to determine the most effective oral hygiene methods for individuals receiving orthodontic treatment.

DETAILED DESCRIPTION:
Because orthodontic appliances cause food retention, a good level of oral hygiene is needed to maintain dental health. Inadequate tooth brushing can lead to gingival diseases on periodontal tissue, cavities and white lesions on tooth enamel. Antimicrobial agents and fluoride products are useful but it cannot replace the mechanical removal of plaque. Because the mechanical plaque control is still considered the most important oral hygiene tool during orthodontic treatment.

In the literature, it has been reported that the motivation to maintain oral hygiene during the orthodontic fixed treatment phase has a very positive effect on periodontal health, and in the same studies, plaque index scores increased over time in control groups that were not given repeated oral treatment. If patients are not given repeated and regular oral hygiene motivation in every session in the clinical routine, gum health may deteriorate. More invasive methods may be required to correct this condition. Because poor oral hygiene, if left unchecked, can compromise the outcome of orthodontic treatment.

When performing manual tooth brushing, the modified Bass technique (MBT) is often recommended to provide optimum plaque reduction by protecting oral tissues from mechanical irritation. The problem with this brushing technique is that it consists of a complex sequence of movements. First of all, the toothbrush should be positioned at a 45° angle to the gingival edge. Secondly, the brush should be moved back and forth with small horizontal vibrations. Thirdly, debris must be removed by sweeping the brush towards the occlusal face in a vertical motion (upward in the lower jaw, downwards in the upper jaw). This sequence of movements requires dexterity and attention to technique. Brushing demonstration techniques or sequences have been developed through a brochure, a model, or video.

ELIGIBILITY:
Inclusion Criteria:

* The patient with orthodontic attachments at least 4 months
* with permanent dentition

Exclusion Criteria:

* impacted or atypically erupted teeth
* with prosthetic restorations such as crowns or implants
* open bite
* deep bite
* crowding more than 7 mm or polydiastema cases
* Individuals diagnosed with periodontitis
* ndividuals with cleft lip and palate or other craniofacial anomalies

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
The Turesky modified index | Baseline, 1st month, 3rd month
  The Turesky modified index, plaque on the buccal and lingual surfaces of all teeth. TMQHI scores were recorded as follows:
  0, no dental plaque present,
  1. isolated areas of dental plaque,
  2. A thin dental plaque tape of ≤1 mm,
  3. dental plaque covered up to 1/3 of the tooth surface,
  4. dental plaque covered between 1/3 and 2/3 of the tooth surface,
  5. dental plaque covers ≥2/3 of the tooth surface.
Orthodontic plaque index | Baseline, 1st month, 3rd month
  Score 0: No plaque accumulation Score 1: There is plaque accumulation covering one side of the bracket base Score 2: There is plaque accumulation covering two sides of the bracket base Score 3: There is plaque accumulation covering three sides of the bracket base Score 4: There is plaque accumulation covering all four sides of the bracket base. and/or the presence of gingival inflammation

SECONDARY OUTCOMES:
Gingival Index | Baseline, 1st month, 3rd month
  Score 0: Healthy gingiva, Score 1: Gingival characterised by mild inflammation, mild discolouration, mild oedema, no bleeding on probing, Score 2: Moderate inflammation, gingiva shiny, red and oedematous. There is bleeding on probing, Score 3: Severe inflammation, marked redness and oedema. There is a tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin TUNCA, PhD, Principal Investigator — Yuzuncu Yil University; Dicle ALTINDAL, DDS, Study Director — Yuzuncu Yil University; Nihal FAHRZADEH, PhD, Study Chair — Yuzuncu Yil University; Murat Tunca, PhD, Study Chair — Yuzuncu Yil University
Locations (1):
- Yasemin TUNCA, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cozzani M, Ragazzini G, Delucchi A, Mutinelli S, Barreca C, Rinchuse DJ, Servetto R, Piras V. Oral hygiene compliance in orthodontic patients: a randomized controlled study on the effects of a post-treatment communication. Prog Orthod. 2016 Dec;17(1):41. doi: 10.1186/s40510-016-0154-9. Epub 2016 Dec 19. PMID 27891568
- [Result] Renton-Harper P, Addy M, Newcombe RG. Video instruction to establish a panel of experts to compare tooth cleaning by 4 electric toothbrushes. J Clin Periodontol. 2001 Oct;28(10):917-22. doi: 10.1034/j.1600-051x.2001.028010917.x. PMID 11686809
- [Result] Diamanti-Kipioti A, Gusberti FA, Lang NP. Clinical and microbiological effects of fixed orthodontic appliances. J Clin Periodontol. 1987 Jul;14(6):326-33. doi: 10.1111/j.1600-051x.1987.tb00979.x. PMID 3509967